CLINICAL TRIAL: NCT02066649
Title: A Phase 3 Study of Carvedilol vs Variceal Band Ligation vs Combination Therapy for Primary Prophylaxis of Variceal Bleeding
Brief Title: Carvedilol vs Band Ligation vs Combination Therapy for Primary Prophylaxis of Variceal Bleeding
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: We need to revise and redesign the study
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Nikolaos T. Pyrsopoulos, MD, PhD, MBA, FACP, AGAF, FAASLD, F, Professor of Medicine and Chief of Gastroenterology & Hepatology, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2013003729
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Portal Hypertension Related to Cirrhosis
Keywords: portal hypertension; esophageal varices; variceal bleed; carvedilol; variceal band ligation
MeSH Terms: conditions — Hypertension, Portal; Esophageal and Gastric Varices | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Carvedilol (Active Comparator): Initiating patient on carvedilol after diagnosis of varices made on endoscopy
  Interventions: Drug: Carvedilol
- Variceal Band Ligation (Active Comparator): performing variceal band ligation during endoscopy on patient after diagnosis of esophageal varices made on endoscopy
  Interventions: Procedure: Variceal band ligation
- Combination Group (Carvedilol + Variceal band ligation) (Active Comparator): once patient has confirmed large esophageal varices on endoscopy, he/she will be started on carvedilol (post-procedure) in addition to having variceal band ligation performed during endoscopy
  Interventions: Drug: Carvedilol; Procedure: Variceal band ligation

INTERVENTIONS:
Drug: Carvedilol — Administering carvedilol to patients diagnosed with large varices on endoscopy
  Other Names: Coreg
  Arms: Carvedilol; Combination Group (Carvedilol + Variceal band ligation)
Procedure: Variceal band ligation — Performing variceal band ligation during endoscopy after diagnosis of large varices on endoscopy
  Arms: Combination Group (Carvedilol + Variceal band ligation); Variceal Band Ligation

SUMMARY:
Subjects will be those individuals greater than 18 years of age with a diagnosis of cirrhosis undergoing screening for esophageal varices. Eligible subjects will have a diagnosis of cirrhosis and esophageal varices (graded as medium or large) with no prior history of variceal bleeding. The diagnosis of cirrhosis will be based on clinical, radiologic, and/or laboratory data. Patients will be randomly assigned using electronic medical records to one of three treatment arms after screening esophagogastroduodenoscopy (EGD) has been performed and large varices are identified. Primary outcome of the study will be the incidence of variceal bleeding in patients receiving one of the following therapies for primary prophylaxis of variceal bleeding: carvedilol, variceal band ligation (VBL), or both carvedilol and VBL.

DETAILED DESCRIPTION:
Inclusion criteria for the study will be an individual > 18 years old with a diagnosis of cirrhosis (either by history, serology or imaging), with medium or large esophageal varices on variceal screening esophagogastroduodenoscopy (EGD), and no prior history of gastrointestinal (GI) bleeding, as related to portal hypertension. Exclusion criteria will be the following: pregnant females; patients on beta blockers or nitrates for any underlying condition; allergies to carvedilol; mean arterial pressure < 55 mm Hg or pulse < 55 beats per minute at baseline; presence of hepatocellular carcinoma; presence of portal vein thrombosis; patients with severe, uncontrolled respiratory disease (asthma, COPD); patients with complete heart block or other significant arrhythmias; those with significant renal disease (CKD stage III or higher); patients who are unable to provide consent; and patients who in the opinion of the principal investigator are not suitable for participation in the trial.

Patients will be randomized to one of the following three treatment groups: (1) carvedilol group, (2) variceal band ligation and (3) combination therapy (carvedilol plus variceal band ligation). Since the standard of care at University Hospital is use of beta blocker medications, the carvedilol group will serve as the control group.

After consent has been obtained for the EGD and research study and patients have met the non-endoscopic inclusion and exclusion criteria mentioned above, they will undergo a screening EGD to look for varices. Varices will be graded by the 2-group classification system of "small" and "large". Varices are graded as large if > 5mm and small if < 5mm in size. A biopsy forceps will be inserted through the biopsy channel of the gastroscope and opened. An open biopsy forceps measures approximately 5mm in diameter. This will be used to measure the size of the varices and will be confirmed by two physicians. If a patient is found to have small esophageal varices, they will be excluded from the study and managed as per the standard of care. Once a patient has been identified in having large esophageal varices, he or she will undergo randomization during that initial endoscopy. A random number generator will be used to randomize the patient into one of the three treatment groups described above. If a patient is randomized to the carvedilol group, the endoscopic procedure will be terminated and the patient will be given a prescription for carvedilol at the time of discharge. He or she will then be followed up in our Gastroenterology clinics in a regular fashion where medication can be titrated and symptoms can be assessed. If a patient is randomized to the variceal band ligation group, the patient will undergo banding of the esophageal varices with a Wilson-Cook multi-banding device. He/she will be started on a proton-pump inhibitor post-procedure to minimize the risk of post-banding ulcers, a known complication of variceal banding. Once the patient has been treated with VBL, this procedure will be scheduled and repeated every two weeks until the obliteration of varices (ie once varices cannot be detected on endoscopy). The first surveillance EGD after obliteration will then be performed 1-3 months after obliteration and then every 6 months to check for variceal recurrence. If a patient is randomized to the combination group, the patient will undergo the banding protocol described above. The patient will then be given a prescription for carvedilol and a proton-pump inhibitor on discharge and followed in our clinics as scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the study will be an individual > 18 years old with a diagnosis of cirrhosis (either by history, serology or imaging), with medium or large esophageal varices on variceal screening esophagogastroduodenoscopy (EGD), and no prior history of gastrointestinal (GI) bleeding, as related to portal hypertension

Exclusion Criteria:

* Exclusion criteria will be the following: pregnant females; patients on beta blockers or nitrates for any underlying condition; allergies to carvedilol; mean arterial pressure < 55 mm Hg or pulse < 55 beats per minute at baseline; presence of hepatocellular carcinoma; presence of portal vein thrombosis; patients with severe, uncontrolled respiratory disease (asthma, COPD); patients with complete heart block or other significant arrhythmias; those with significant renal disease (CKD stage III or higher); patients who are unable to provide consent; and patients who in the opinion of the principal investigator are not suitable for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of first variceal bleed | within 2 year follow-up period

SECONDARY OUTCOMES:
Bleed-related mortality | within 2-year follow-up period
Overall mortality | Within 2 year follow-up period
Recurrence of varices | within 2 year follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: NIKOLAOS T PYRSOPOULOS, MD, Principal Investigator — RUTGERS - NJMS- DEPARTMENT OF MEDICINE
Locations (1):
- Rutgers NJ Medical School, Newark, New Jersey, United States

REFERENCES:
- [Background] Garcia-Tsao G, Sanyal AJ, Grace ND, Carey W; Practice Guidelines Committee of the American Association for the Study of Liver Diseases; Practice Parameters Committee of the American College of Gastroenterology. Prevention and management of gastroesophageal varices and variceal hemorrhage in cirrhosis. Hepatology. 2007 Sep;46(3):922-38. doi: 10.1002/hep.21907. No abstract available. PMID 17879356